CLINICAL TRIAL: NCT02354495
Title: Individualized Metabolic Assessment and Nutritional Optimization in Children With Chronic Respiratory Insufficiency on Ventilatory Support at Home
Brief Title: Individualized Metabolic Assessment and Nutritional Optimization in Children With Chronic Respiratory Insufficiency
Acronym: NutriCAPE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Nilesh M. Mehta, Associate Professor in Anesthesia, Critical Care, Boston Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: P00004109
Record Dates: First submitted 2015-01-29; First posted 2015-02-03 (Estimated); Last update posted 2016-01-27 (Estimated); Status verified 2016-01

CONDITIONS: Nutrition
Keywords: Indirect calorimetry; Protein; Mechanical ventilation; Respiratory failure
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Diet intervention arm (Experimental): Individualized diet prescription following food record, indirect calorimetry (for energy requirement) and body composition assessments. repeat assessments after 12 weeks on interventional diet.
  Interventions: Dietary Supplement: Changes in energy and protein intake

INTERVENTIONS:
Dietary Supplement: Changes in energy and protein intake — Energy intake will be based on accurate measurements of energy expenditure. Protein intake will be matched to age-based recommended values if necessary.

SUMMARY:
The investigators aim to examine the feasibility of individualized diet intervention in children dependent on long-term mechanical ventilator support at home. The investigators will use a multidisciplinary model that will allow for diet modification based on comprehensive nutrition, metabolic and respiratory assessments performed in the subjects' home. the impact of this intervention (for 12 weeks) on body composition and respiratory variables will be assessed.

DETAILED DESCRIPTION:
A strategy of individualized diet intervention and its impact on respiratory and nutritional outcomes in children on long-term mechanical ventilation has not been previously evaluated.

The investigators' objective is to assess the feasibility of individualized diet intervention in children dependent on long-term mechanical ventilator support using a multidisciplinary model. The investigators will optimize energy intake (based on indirect calorimetric measurement) and protein intake (based on recommended intake values) in this group. The subjects will be administered the modified diet for 12 weeks, and a comprehensive nutrition, metabolic and respiratory assessment will be performed before and after intervention, in the subjects' home. The investigators will examine the effect of individualized diet optimization on nutritional status, body composition, CO2 production (VCO2) and minute ventilation (MV).

The investigators hypothesize that optimizing energy and protein intake would be associated with improved nutritional status, particularly increment in LBM, and decrease in VCO2 and MV. If nutritional optimization is associated with positive outcomes in our study cohort, this concept could be generalized to a wider patient population with respiratory insufficiency.

ELIGIBILITY:
Inclusion Criteria:

- Children aged 1 month to 17 years will be included if they were dependent on at least 12 hours of mechanical ventilation per day via a cuffed tracheostomy tube, with a fractional oxygen requirement (FiO2) less than 0.6, and a leak less than 10% around the cuff at the time of data collection

Exclusion Criteria:

-Intercurrent illness such as fever, seizures and/or infectious disease in the 24 hours preceding the study, and/or respiratory decompensation requiring an increase in ventilator settings of >20% from baseline in the 72 hours preceding the study

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 16 (Actual)
Dates: Start 2013-08; Primary Completion 2014-08 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Lean body mass | 12 weeks
  change in LBM after 12 weeks of modified diet
Carbon dioxide production (VCO2) | 12 weeks
  Change in VCO2 (ml/min) after 12 weeks on modified diet
Minute ventilation (L/min) | 12 weeks
  Change in minute ventilation (L/min) after 12 weeks on modified diet

REFERENCES:
- [Background] Martinez EE, Smallwood CD, Bechard LJ, Graham RJ, Mehta NM. Metabolic assessment and individualized nutrition in children dependent on mechanical ventilation at home. J Pediatr. 2015 Feb;166(2):350-7. doi: 10.1016/j.jpeds.2014.09.036. Epub 2014 Oct 25. PMID 25444009